CLINICAL TRIAL: NCT01176903
Title: Randomized, Double-blind, Placebo-controlled, Cross-over Study to Investigate the Bronchodilator Efficacy and Safety After Single and Repeated Administrations of Different Doses of Glycopyrrolate Via pMDI in Moderate to Severe COPD Patients.
Brief Title: Safety and Efficacy Study of Glyco pMDI After Single and Repeated Administration
Acronym: GLY2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0916-PR-0032; 2010-018668-18 (EudraCT Number)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Glyco SD1 (Experimental): Single administration of Glyco pMDI dose level 1
  Interventions: Drug: Glycopyrrolate
- Glyco SD2 (Experimental): Single administration of Glyco pMDI dose level 2
  Interventions: Drug: Glycopyrrolate
- Glyco SD3 (Experimental): Single administration of Glyco pMDI dose level 3
  Interventions: Drug: Glycopyrrolate
- Glyco SD4 (Experimental): Single administration of Glyco pMDI dose level 4
  Interventions: Drug: Glycopyrrolate
- Glyco SD5 (Experimental): Single administration of Glyco pMDI dose level 5
  Interventions: Drug: Glycopyrrolate
- Placebo SP (Placebo Comparator): Single administration of Placebo pMDI
  Interventions: Drug: placebo
- Glyco MD1 (Experimental): Multiple administration of Glyco pMDI dose level 1
  Interventions: Drug: Glycopyrrolate
- Glyco MD2 (Experimental): Multiple administration of Glyco pMDI dose level 2
  Interventions: Drug: Glycopyrrolate
- Glyco MD3 (Experimental): Multiple administration of Glyco pMDI dose level 3
  Interventions: Drug: Glycopyrrolate
- Placebo MP (Placebo Comparator): Multiple administration of placebo pMDI
  Interventions: Drug: placebo
- Tiotropium (Active Comparator): Multiple administration of tiotropium
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Glycopyrrolate — pressurized metered dose inhaler
  Other Names: CHF 5259
  Arms: Glyco MD1; Glyco MD2; Glyco MD3; Glyco SD1; Glyco SD2; Glyco SD3; Glyco SD4; Glyco SD5
Drug: Tiotropium — inhalation powder, hard capsule
  Other Names: Spiriva
  Arms: Tiotropium
Drug: placebo — pressurized metered dose inhaler
  Arms: Placebo MP; Placebo SP

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of Glycopyrrolate as pMDI after single and repeated administration.

DETAILED DESCRIPTION:
The study is divided into two parts:

- Part 1 will be conducted according to a single-centre, randomized, double-blind, placebo-controlled, single-dose escalation, alternating crossover design in two groups of COPD patients.

Treatments to be administered on Part 1 (SD1, SD2, SD3, SD4, SD5, SP). The primary objective of Part 1 is the evaluation of the safety and tolerability of Glyco after single administration.

- Part 2 will be conducted according to a single-centre, randomized, double-blind, placebo-controlled, 4-period, 4-treatment, repeated dose cross-over design followed by an open-label extension period with tiotropium.

Treatments administered on Part 2 (MD1, MD2, MD3, MP, Tiotropium). On the last treatment day in the morning, Formoterol 12 µg will be administered to all patients on top of placebo or Glyco or Tiotropium.

The primary objective of Part 2 is the evaluation of the efficacy of Glyco after repeated administration.

Part 2 will start after a safety review of the results obtained from Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Males and females patients aged 40-75 years;
* Written informed consent obtained;
* Diagnosis of moderate-severe COPD, according to the GOLD guidelines;
* Current or ex-smokers with a smoking history of ≥ 10 pack-years
* Post bronchodilator FEV1 between 40% and 80% predicted values (40% ≤ FEV1 < 80%), documented at screening visit ;
* Post bronchodilator FEV1/Forced Vital Capacity (FEV1/FVC) ≤ 0.70 (absolute value) documented at screening visit;
* Airway reversibility of at least 100 mL within 30 to 45 minutes after inhalation of ipratropium 80µg.

Exclusion Criteria:

* History of chronic or seasonal allergy
* Blood eosinophil count above 600 per µl
* Clinically relevant findings on physical examination laboratory and ECG parameters at screening
* Occurrence of clinically relevant abnormalities in the 24-h Holter ECG recording at screening;
* Significant disease not related to COPD (eg. Myocardial infarction, stroke within the preceding 6 months);
* Respiratory tract infection (including upper tract) 4 weeks prior to study entry requiring changing treatment;
* Patients requiring oxygen therapy on a daily basis for chronic hypoxemia;
* History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency, or any other significant lung disease which is considered to be clinically significant by the investigator.
* Intolerance/hypersensitivity or any contra-indication to treatment with M3 Antagonist or any of the excipients contained in the formulations used in the study.
* History of alcohol or substance abuse that in the opinion of the Investigator may be of clinical significance.
* Patients treated with slow-release oral or parental corticosteroids 8 weeks prior to Screening Visit.
* Patients treated with tiotropium in the 10 days prior to the Screening Visit;
* Pregnant or lactating women and female or male subjects not willing to use an acceptable method of contraception.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 24 hours after single administration
  Adverse events, vital signs, ECG parameters, 24-hours ECG holter recording, clinical laboratory abnormalities.
  This primary outcome is for the Part 1 of the study.
Lung function (trough FEV1) | 12 hours post dose after repeated administration
  This primary variable is for the Part 2 of the study.

SECONDARY OUTCOMES:
Lung function | up to 24 hours post dose
  for Part 1 of the study
Lung function (other parameters) | up to 12 hours after repated administration
  for Part 2 of the study
Body plethysmography | up tp 12 hours after repeated administration
  for Part 2 of the study
Pharmacokinetics | up to 12 hours after single and repeated administration
  Pharmacokinetics in plasma and urine. For Part 2 of the study.
Safety | up to 12 hours after single and repeated administration
  Adverse events, Vital signs, ECG parameters, 24-hour ECG holter recording. For Part 2 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit Ltd
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom

REFERENCES:
- [Result] Singh D, Scuri M, Collarini S, Vezzoli S, Mariotti F, Muraro A, Acerbi D. Bronchodilator efficacy of extrafine glycopyrronium bromide: the Glyco 2 study. Int J Chron Obstruct Pulmon Dis. 2017 Jul 7;12:2001-2014. doi: 10.2147/COPD.S137659. eCollection 2017. PMID 28744115
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-018668-18
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-0916-PR-0032.pdf